CLINICAL TRIAL: NCT06972043
Title: Development and Testing of an AI-Assisted Smart Interactive Healthcare Robot Program
Brief Title: AI-Assisted Smart Interactive Healthcare Robot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202410046RINE
Record Dates: First submitted 2025-04-07; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Nursing; Artificial Intelligence (AI); Deep Learning; Mechine Learning
Keywords: Nursing; Artificial Intelligence (AI); Medical Science and Technology

STUDY DESIGN:
Intervention Model Description: Since the robot will interact with patients or caregivers during its operation in the ward, in addition to the nursing staff completing the informed consent form, patients or caregivers will also be required to fill out a consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Other): The functions performed by the robot include guiding patients through unit-specific locations for environmental orientation and equipment usage instructions, playing educational videos related to care, reminding patients of important examination precautions, providing health education on specimen collection, and delivering responses through an expert-developed medical Q&A system.
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — The functions performed by the robot include guiding patients through unit-specific locations for environmental orientation and equipment usage instructions, playing educational videos related to care, reminding patients of important examination precautions, providing health education on specimen collection, and delivering responses through an expert-developed medical Q&A system.

SUMMARY:
To address workforce shortages and increasing workloads in nursing, technological solutions and AI-powered robots for ward navigation have been introduced. However, limitations remain in their application to clinical care. This study aims to develop and test a programming framework for an AI-assisted nursing care robot ("E-Nursing Assistant") to reduce nurses' workload and improve the efficiency and quality of care.

DETAILED DESCRIPTION:
In response to the challenges of workforce shortages and heavy workloads in the nursing field, clinical nursing practices are gradually integrating technological assistance, including the use of mobile phones to scan QR codes for viewing instructional videos and the introduction of robots with Artificial Intelligence (AI) technology for ward navigation. However, there are still several limitations to these technological applications in the nursing care process. Therefore, this study aims to develop and test the programming framework for an AI-assisted nursing care robot ("E-Nursing Assistant"). The goal is to reduce the workload of nursing staff and significantly improve the efficiency and quality of nursing work. The "E-Nursing Assistant" will be implemented in the ward to measure the nursing staff's workload, the time and frequency spent on specific nursing tasks, and to conduct interviews to gather their feedback.

ELIGIBILITY:
1. Nurse

   Inclusion Criteria:
   * Aged 18 years or older.
   * Currently employed as a ward nurse.

   Exclusion Criteria:
   * Nurses who do not actively participate in ward care, such as nursing unit supervisors.
2. Patients/Caregivers

Inclusion Criteria:

* Aged 18 years or older.
* Willing to accept the "E-Nursing Assistant" intervention for care tasks that do not involve patient safety.

Exclusion Criteria:

* Patients or caregivers who are unconscious or unable to communicate verbally or in writing to complete the research interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Workload-related stress in nursing staff | It will be measured pre-intervention and immediately after the intervention.
  The investigators utilized the Nurse Stress Checklist Chinese version translated by Taiwanese scholars in 1996. The scale consists of four factors: "Personal Response," "Work Concerns," "Job Competence," and "Inability to Complete Personal Tasks." It contains a total of 43 items, each rated on a 9-point Likert scale (0 = not at all, 1 = not close, 8 = very close), with higher scores indicating greater levels of work-related stress.

SECONDARY OUTCOMES:
System Usability | It will be measured immediately after the intervention.
  The investigators used the System Usability Scale (SUS) developed by scholar Brooke. The scale consists of 10 items, scored on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Odd-numbered items are positively worded, and the raw score for each item is subtracted by 1 to obtain the item score. Even-numbered items are reverse scored, with the item score calculated as 5 minus the raw score. The scores for all items are summed, and the total is then multiplied by 2.5 to obtain the overall SUS score, which ranges from 0 to 100. Higher scores indicate greater satisfaction with the system.
Number of patients served and time spent on various nursing tasks | It will be measured pre-intervention and during the intervention
  A self-designed table will be used to list common and repetitive nursing tasks in the ward in detail. These tasks include: ward orientation (e.g., nursing station), instructions for using ward equipment (e.g., patient beds, call bells), patient fall prevention education, reminders for various examinations (e.g., urination), health education for specimen collection (e.g., blood, urine), discharge instructions, and answering common questions from patients after viewing nursing care instructional videos. Each task will include spaces to record the number of patients served and time spent. Initially, an audio recorder will be used to measure the time, after which the researchers will calculate the start and end times, as well as any interruptions during the process, and fill in the table accordingly.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided